CLINICAL TRIAL: NCT01153620
Title: Randomized, Double-blind, Controlled Clinical Trial on the Antiseptic Efficacy and Tolerability of Lavasept® 0.04% on Acute Traumatic Wounds
Brief Title: The Antiseptic Efficacy and Tolerability of Lavasept® 0.04% on Acute Traumatic Wounds
Acronym: Lavasept 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Ltd. Centre of Excellence Infection Control (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPM-CIC-G-H-0901
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Wounds
Keywords: Acute traumatic wounds
MeSH Terms: conditions — Wounds and Injuries | interventions — Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ringer's Solution (Placebo Comparator)
  Interventions: Other: Ringer's Solution
- Lavasept 0.04% (Active Comparator)
  Interventions: Drug: Lavasept 0.04%

INTERVENTIONS:
Drug: Lavasept 0.04% — Method of Administration A sterile compress will be saturated with Lavasept® 0.04% / Ringers' solution and placed on the wound.
  Dosage Lavasept® 0.04% 50 ml 50ml or as much needed to completely saturate the compress.
  Treatment Duration 60 minutes
  Arms: Lavasept 0.04%
Other: Ringer's Solution — Method of Administration A sterile compress will be saturated with Lavasept® 0.04% / Ringers' solution and placed on the wound.
  Dosage Ringers' solution 50ml or as much needed to completely saturate the compress. Treatment Duration 60 minutes
  Arms: Ringer's Solution

SUMMARY:
The primary objective of the study is to assess the antiseptic efficacy of Lavasept 0.04% when used as an antiseptic agent and to compare these with Ringers' solution in patients with acute traumatic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute traumatic cut, crush, abrasion, bite or stab wounds Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the Institutional Ethics Committee (IEC) prior to all evaluations
* Wounds that are a minimum of approximately 4 cm2 in size
* Ability to read and understand the German patient information sheet and informed consent form

Exclusion Criteria:

* < 18 years of age
* Pregnancy
* Immunosuppression
* Wounds caused by a burn
* Wounds that require treatment of hyaline cartilage, the central nervous system, peritoneum, meningae, inner / middle ear or inner eye
* Simultaneous participation in another clinical trial
* Wounds that require immediate surgical or medical treatment as well patients who are critically ill
* Patient with a known allergy to the active agent or any of the excipients
* Wounds that are >3 cm in depth
* Wounds that have not received medical treatment for ≥6 hours
* Heavily bleeding wounds
* Open fractures, joints or tendons
* Wounds of the face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Peter Simmen, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Emergency roon in University Hospital
Period: Overall Study
Arm/Group | Ringer's Solution | Lavasept 0.04%
Started | 30 | 30 (30 patients (31 wounds))
Completed | 30 | 30 (30 patients (31 wounds))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ringer's Solution | Lavasept 0.04% | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 8 | 9 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 47.63 (24.487) | 47.68 (23.019) | 47.66 (23.553)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 23 | 27 | 50
Region of Enrollment [Number; unit: participants]
  Switzerland | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Reduction (log10) in Colony Forming Units
Description: Comparison of the log10 reduction in CFU after 60 minutes of treatment application.
Time Frame: 60 minutes
Population: ITT population: comprising all wounds having received the study treatment for any duration (n=61).
Measure: Mean (Standard Deviation); unit: log 10 Colony Forming Units
Units Other Than Participants: wounds
Groups:
- Lavasept 0.04%; Ringer's Solution: Reduction in log 10 Colony Forming Units after 60 minutes of treatment
Arm/Group | Lavasept 0.04% | Ringer's Solution
Number analyzed (Participants) | 30 | 30
Number analyzed (wounds) | 31 | 30
log 10 Colony Forming Units | 0.734 (1.00) | -0.06 (0.85)
Statistical Analysis 1: Comparison: Lavasept 0.04% vs Ringer's Solution; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Local Tolerability: Pruritis Burning
Description: Local tolerability after 60 minutes of treatment application.
Time Frame: 60 minutes
Reporting Status: Not Posted

3. Secondary Outcome: Reduction in CFU
Description: Comparison of the percentage reduction in CFU after 15, 30 and 60 minutes of treatment application
Time Frame: 15 minutes, 30 minutes and 60 minutes
Reporting Status: Not Posted

4. Secondary Outcome: Comparison of the Percentage of Patients With Target Wounds <50 CFU
Description: Comparison of the percentage of patients with target wounds <50 CFU after 60 minutes of treatment application
Time Frame: 60 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ringer's Solution | Lavasept 0.04%
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less